CLINICAL TRIAL: NCT03738800
Title: A Phase 2 Randomized, Multicenter, Double-blind, Vehicle Controlled, 90-Day, Safety, Efficacy & Systemic Exposure Study of Trifarotene (CD5789) Cream HE1 in Adults and Adolescents With Autosomal Recessive Ichthyosis With Lamellar Scale
Brief Title: A Safety, Efficacy and Systemic Exposure Study of CD5789 Cream in Adults and Adolescents With Lamellar Ichthyosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-ICH-001
Record Dates: First submitted 2018-10-24; First posted 2018-11-13 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-02

CONDITIONS: Lamellar Ichthyosis
MeSH Terms: conditions — Ichthyosis, Lamellar | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CD5789 Cream 200 µg/g (Experimental): CD5789 200 µg/g, topical, 50g
  Interventions: Drug: CD5789 Cream 200 µg/g
- CD5789 Cream 100 µg/g (Experimental): CD5789 100 µg/g, topical, 50g
  Interventions: Drug: CD5789 Cream 100 µg/g
- CD5789 Cream Vehicle (Placebo Comparator): CD5789 Cream Vehicle, topical, 50g
  Interventions: Drug: CD5789 Cream Vehicle

INTERVENTIONS:
Drug: CD5789 Cream 200 µg/g — A fixed dose (determined at Visit 1) of 200 µg/g applied topically twice weekly to up to 90% BSA
  Arms: CD5789 Cream 200 µg/g
Drug: CD5789 Cream 100 µg/g — A fixed dose (determined at Visit 1) of 100 µg/g applied topically twice weekly to up to 90% BSA
  Arms: CD5789 Cream 100 µg/g
Drug: CD5789 Cream Vehicle — A fixed dose (determined at Visit 1) applied topically twice weekly, up to 36 g per dose up to 90% BSA
  Arms: CD5789 Cream Vehicle

SUMMARY:
This is a phase 2 randomized, multi-center, double-blind, vehicle controlled, 90 day, safety, efficacy, and systemic exposure study followed by a 90 day open-label extension of trifarotene cream in adults and adolescents with autosomal recessive ichthyosis with lamellar scale.

DETAILED DESCRIPTION:
This is a 2-cohort, multicenter study in subjects with moderate to severe LI. Adults (Cohort A) and adults and adolescents (Cohort B) will be randomized in a double-blind fashion to 1 of 2 doses of active or vehicle and treated twice weekly for 90 days. Subjects who complete the randomized, double-blind portion of the study will be eligible to enter a 90 day, open-label extension study.

Approximately 15 adults (≥18 years old) will be randomized into the first cohort of subjects (Cohort A) in a 1:1:1 ratio and treated twice weekly for up to 90 days. If no safety issues are identified, both adults and adolescents (ages 12-17 years, inclusive) will be allowed to enroll in Cohort B. Subjects in Cohort B will be randomized 1:1:1 and treated twice weekly for up to 90 days in the same manner as subjects in Cohort A.

All subjects who complete 90 days of double-blind study treatment will be eligible to enroll in a 90 open-label extension. Subjects in the open-label extension will receive active twice weekly for up to 90 days.

ELIGIBILITY:
1. For Cohort A: subject is ≥18 years old; for Cohort B: subject is ≥12 years old.
2. Subject has known diagnosis of LI.
3. Subject has moderate to severe (IGA 3-4) LI on the IGA of LI severity.
4. Subject has signed an ICF at Screening before any investigational procedures. Subjects <18 years of age (or Age of Majority) must sign an assent form in conjunction with an ICF signed by the parent/legal representative.
5. Subject who is participating in optional photography has signed a photography ICF.
6. Subject who is participating in the optional PK substudy has signed a PK ICF. Minors, in the event of their reaching majority during the study, should be capable of giving consent to take part in the PK substudy.
7. Subject is not of childbearing potential, who is postmenopausal (absence of menstrual bleeding for 1 year before Baseline, without any other medical reason), or has documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy. For individuals with permanent infertility due to an alternate medical cause other than the above, (e.g., Mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

   OR
   * Subject is a woman of childbearing potential (WOCBP), i.e., a female ≥12 years of age (regardless of whether they have experienced/reported menarche), or a male subject with sexual partners capable of reproduction who agrees to use 2 effective forms of contraception during the study and for at least 1 month after the last study drug application. The 2 authorized forms of contraception are condom used with 1 of the following methods of contraception:
   * bilateral tubal ligation
   * combined oral contraceptives (estrogens and progesterone), vaginal ring, or implanted or injectable hormonal contraceptives with a stable dose for at least 1 month before Baseline; hormonal contraceptives must inhibit ovulation
   * intrauterine device (IUD) inserted at least 1 month before Baseline OR Agrees to abstain from heterosexual intercourse during study participation and for 1 month after the last application of study drug and to use a highly effective contraceptive as backup if he or she becomes sexually active during the study. Abstinence is only acceptable if this is the subject's usual lifestyle. Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception.

   AND Male subjects may not donate sperm during the study and for at least 1 month after the last study drug application.

   Note: Female subjects who are premenstrual at screening should nonetheless follow the pregnancy testing schedule for WOCBP even if they abstain from sexual intercourse while in the study and for at least 1 month after the last study drug application.
8. Women of childbearing potential must be nonlactating and have negative pregnancy test results at Screening (serum) and on Day 1 before study drug administration (urine).
9. Subject is reliable and capable of adhering to the protocol and visit schedule, in the investigator's judgment, and has signed informed consent/assent, as applicable.
10. Subject is taking no more than 3500 IU/day Vitamin A (e.g., as in a multivitamin).

Exclusion criteria:

1. Subject has any variant of ichthyosis other than LI or another disorder of keratinization, including syndromic ichthyoses.
2. Subject has current moderate or severe stinging/burning at Screening.
3. Subject has an ongoing cutaneous infection or any other significant concomitant skin disease (other than the LI) which, in the investigator's opinion, may interfere with the study assessments.
4. Subject with fasting triglycerides >200 mg/dL or >2.25 mmol/L and/or total cholesterol >250 mg/dL or >6.5 mmol/L. Subjects whose triglycerides and/or total cholesterol are within normal limits with a stable dose of lipid-lowering agents for at least 6 months may be included.
5. Subject was previously treated with trifarotene/CD5789 in an acne or ichthyosis study.
6. Subject has any other significant concomitant disease, or poorly controlled medical condition other than LI that in the investigator's opinion may put him or her at risk if he or she takes part in the study, and/or that may interfere with the study assessments.
7. Subject has a medical condition that potentially alters bone metabolism (e.g., osteoporosis, thyroid dysfunction, Cushing syndrome, Crohn's disease, or ulcerative colitis). Subjects with hypothyroidism who are on a stable dose of thyroid hormone replacement therapy and whose thyroid-stimulating hormone (TSH) is normal may be included
8. Subject is being treated for major depression disorder and/or has a history of major depression or suicide attempt requiring hospitalization, medications, and close psychiatric surveillance to prevent suicide attempts.
9. Subject with positive serology for hepatitis B surface antigen, hepatitis C, or are known to be HIV positive or to have AIDS at Screening.
10. Subject with any of the following laboratory values at Screening:

    1. Aspartate aminotransferase or alanine aminotransferase >1.5 × upper limit of normal defined by the laboratory
    2. Total bilirubin >1.25 × ULN at Screening. Subjects with known Gilbert's syndrome may be included with total bilirubin >1.25 × ULN
    3. Hemoglobin <12.5 g/dL for men and <11.5 g/dL for women
    4. Platelets <150 × 109/L or >400 × 109/L.
11. Subject has any clinically other significant abnormal laboratory value (hematology, chemistry, or urinalysis) at Screening that, in the investigator's opinion, may put the subject at risk if he or she takes part in the study, and/or that may interfere with the study assessments.
12. Subject has had recent systemic malignancy (e.g., within 5 years) with exception of nonmelanoma skin cancer or cervical intraepithelial neoplasia of Grade 1 who are >6 months post-treatment.
13. Subject has a history of long QT syndrome or has clinically significant electrocardiogram (ECG) abnormalities, including clinically significant conduction disorders or significant arrhythmias, or QTcF interval >450 ms.
14. Subject has a known allergy or sensitivity to any of the components of the investigational products.
15. Subject has been exposed to excessive UV radiations on the treated zones within 1 month before Baseline visit or is planning intensive UV exposure during the study (e.g., occupational exposure to the sun, sunbathing, phototherapy, etc.).
16. Subject is inherently sensitive to sunlight.
17. Subject is unable or unwilling to stop use of topical or systemic retinoids.
18. Subject is presumed to be abusing drug or alcohol at Screening or Baseline Visits based on medical history or current clinical symptoms.
19. Subject is participating in another interventional clinical trial.
20. Subject is institutionalized.
21. Subject is in any way related to the sponsor, investigator, or site personnel.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Choate, MD, Principal Investigator — Yale University
Locations (36):
- United States (10):
  - TCR Medical Corporation, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - NorthShore University HealthSystem, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DermAssociates, PC, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Australia (4):
  - Eastern Health Monash University, Box Hill
  - Veracity Clinical Research, Brisbane
  - Royal Children's Hospital, Parkville
  - Premier Specialists Ptd Ltd, Sydney
- The Hospital for Sick Children, Toronto, Canada
- France (3):
  - Dermatologie pédiatrique, Paris
  - CHU Charles Nicolle, Rouen
  - CHU de Toulouse- Hospital Larrey, Toulouse
- Germany (5):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitätsklinkum Frankfurt, Frankfurt
  - Kath. Kinderkrankenhaus Wilhelmstift, Hamburg
  - Ludwig-Maximilians University, Munich
  - Universitatsmedizin Rostock, Rostock
- Tel Aviv Sourasky Mc, Tel Aviv, Israel
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Nino Jesus, Madrid
  - Clinica Universidad de Navarra (Madrid), Madrid
  - Hospital Niño Jesús, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Ukraine (6):
  - Medical Center of Private Enterprise "Dzerkalo", Dnipro
  - Dnipropetrovsk State Hospital of Dermatovenerology, Dnipro
  - Medical Center "Family Medicine Clinic", Dnipro
  - Ternopil Regional Clinical Dermatovenereological Dispensary, Ternopil
  - TDC PE "Asclepius", Uzhhorod
  - Community Institution "Zaporizhzhya Regional Dermatovenereology Clinical Hospital", Zaporizhzhya
- Royal London Hospital Barts Health Nhs Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Treatment Period
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | CD5789 Cream Vehicle
Started | 23 | 21 | 21
Completed | 14 | 18 | 17
Not Completed | 9 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Study Discontinued By Sponsor | 5 | 3 | 3
Not completed — Lack of Efficacy | 2 | 0 | 1
Period: Open Label Extension
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | CD5789 Cream Vehicle
Started | 49 | 0 (Open-label Extemsion (OLE) received trifarotene cream HE1 200 mcg/g twice weekly for 90 days.) | 0 (Open-label Extemsion (OLE) received trifarotene cream HE1 200 mcg/g twice weekly for 90 days.)
Completed | 39 | 0 | 0
Not Completed | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | CD5789 Cream Vehicle | Total
Number analyzed (Participants) | 23 | 21 | 21 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 4 | 1 | 13
  Between 18 and 65 years | 15 | 14 | 19 | 48
  >=65 years | 0 | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (17.08) | 35.1 (20.70) | 31.5 (13.34) | 32.9 (17.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 14 | 41
  Male | 12 | 5 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 17 | 20 | 60
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 4 | 8
  White | 18 | 15 | 13 | 46
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 3 | 1 | 5
5-point Investigator's Global Assessment [IGA] [Mean (Standard Deviation); unit: units on a scale] — 5-point Investigator's Global Assessment [IGA] where 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe)
  units on a scale | 3.5 (0.51) | 3.5 (0.51) | 3.3 (0.48) | 3.4 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects in Each Treatment Group Who Experienced Successful Resolution of LI.
Description: The percentage of subjects in each treatment group who experienced successful resolution of LI where "success" is defined as clear/almost clear on treated areas and at least a 2-grade change from Baseline at Day 90/end-of-treatment (EOT) in the Double-blind Period on the 5-point IGA full body scale.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | CD5789 Cream Vehicle
Number analyzed (Participants) | 15 | 17 | 17
Participants | 0 | 2 | 0

2. Secondary Outcome: Total 16-point Visual Index for Ichthyosis Severity (VIIS)
Description: 5-point Visual Index for Ichthyosis Severity (VIIS) for scaling (overall 16 points) for scaling, i.e. 0-4 points for 4 body areas: chest/abdomen, back, arms and legs) where minimum is 0 and maximum is 16 (e.g. 4 points for each of the four body parts).
  0 (Clear) No scaling
  1. (Almost Clear) Very fine, non-coalescent scales
  2. (Mild) Small and thin, non-coalescent scales
  3. (Moderate) Large and rather thick scales starting to coalesce
  4. (Severe) Very large, adherent, coalescent and very thick scales
Time Frame: 90 Days
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CD5789 Cream 200 µg/g; CD5789 Cream 100 µg/g; Overall Trifarotene Cream (200 µg/g and 100 µg/g); Vehicle Cream: Intent-to-treat population, secondary outcome
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 15 | 17 | 32 | 17
units on a scale | 10.9 (4.24) | 10.9 (3.51) | 10.9 (3.86) | 11.4 (2.94)

3. Secondary Outcome: The Difference in Mean Scores Using Individual Score for Roughness
Description: The amount of roughness of the skin will be measured on a 5-point scale. 0 (Clear) Smooth skin
  1. (Almost Clear) Hardly palpably roughness
  2. (Mild) Mild roughness (fine sand paper-like)
  3. (Moderate) Moderate, coarse roughness (coarse sand paper-like)
  4. (Severe) Very coarse skin (broken cornflakes-like)
Time Frame: 90 Days
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 15 | 17 | 32 | 17
score on a scale | 2.7 (1.10) | 2.7 (0.99) | 2.7 (1.02) | 3.1 (0.78)

4. Secondary Outcome: The Difference in Mean Scores Using Palm Sole Assessment
Description: Thickening of the skin on the palms and soles will be measured on a 5-point scale:
  0 (Clear) No thickening, no roughness, no fissure
  1. (Almost Clear) Only slight thickening, minimal to no roughness, no fissures
  2. (Mild) Some thickening, mild roughness on palpation, few fissures may be present
  3. (Moderate) Substantial and diffuse thickening, coarse roughness on palpation may be present, fissures may be present
  4. (Severe) Very thickened and rough skin, numerous fissures
Time Frame: 90 Days
Population: Intent-to-treat population, secondary endpoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 15 | 17 | 32 | 17
score on a scale | 2.1 (1.06) | 1.6 (1.27) | 1.9 (1.18) | 2.6 (1.06)

5. Secondary Outcome: The Difference in Proportion of Subjects With Presence of Fissures on Palms Between the Active and Vehicle Groups
Description: Fissuring will be assessed by recording the presence or absence of fissures, the number of fissures present, and the pain associated with each fissure. The subject will assess pain associated with fissures as ranging from 0-3 (none, mild, moderate, severe) at day 90 between the active trifarotene cream HE1 and vehicle groups
Time Frame: 90 Days
Population: Intent-to-treat population, secondary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 15 | 16 | 31 | 17
Participants
  Number of participants with Fissures Present at Day 90 | 5 | 4 | 9 | 7
  Number of participants with no fissures present at day 90 | 10 | 12 | 22 | 10

6. Secondary Outcome: Quality of Life Measurement Per Dermatology Life Quality Index (DLQI)
Description: The DLQI, or the Dermatology Quality of Life Index, is a dermatology-specific Quality of Life instrument. It is a simple 10-question validated questionnaire with 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment); higher scores indicate poorer quality of life. Responses collected are on a scale of 0-3 depending on the question relevance to the subject.
  Response (Score) Very much (scored 3) A lot (scored 2) A little (scored 1) Not at all (scored 0) Not relevant (scored 0) A minimum score of 0 and maximum score of 30 is obtained by summing the score of each question. The higher the score, the more quality of life is impaired.
  0-1 = no effect at all on patient's life 2-5 = small effect on patient's life 6-10 = moderate effect on patient's life 11-20 = very large effect on patient's life 21-30 = extremely large effect on patient's life
Time Frame: 90 Days
Population: Intent-to-treat population, secondary endpoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 11 | 16 | 27 | 17
score on a scale | 6.1 (5.22) | 5.9 (5.21) | 6.0 (5.11) | 6.2 (5.78)

7. Secondary Outcome: The Difference in Proportion of Subjects With Presence of Fissures on Soles Between the Active and Vehicle Groups
Description: as for outcome 5
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | Overall Trifarotene Cream (200 µg/g and 100 µg/g) | Vehicle Cream
Number analyzed (Participants) | 15 | 16 | 31 | 17
Participants
  Numer of participants with fissures on soles present at day 90 | 5 | 4 | 9 | 7
  Numer of participants with no fissures on soles present at day 90 | 10 | 12 | 22 | 10

8. Other Pre Specified Outcome: The Difference in Mean Ectropion Scores Between the Active and Vehicle Groups
Description: The Ectropion Severity Score (ESS), is a proven system to be reliable and sensitive to the presence of ectropion and has a maximum score of 8 points (0-8). A higher score indicates a worse ectropion. The score takes the severity of ectropion in terms of lateral and medial apposition, scleral show, conjunctival show, and roundness of the eye into account and gives an indication of the functional aspects involved in ectropion by scoring redness, excess tear film, and the position of the lacrimal punctum A point scale of 0=Nonaffected, 0.5=Emerging, 1= Affected is assigned to 8 observations.
  * Lateral apposition
  * Medial apposition
  * Sceral show
  * Conjunctival show
  * Excess team film
  * Redness of the eye
  * Round canthus
  * Punctum lacrimale
Time Frame: 180 Days
Population: Intent-to-treat population, open label extension
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CD5789 Cream 200 µg/g: Intent-to-treat population, open label extension
Arm/Group | CD5789 Cream 200 µg/g
Number analyzed (Participants) | 38
score on a scale | 2.82 (3.077)

9. Other Pre Specified Outcome: Quality of Life Measurement Per EQ-5D-5L
Description: The EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ visual analog scale (VAS). Descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 5 responses.
  1. no problem
  2. slight problems
  3. moderate problems
  4. severe problems
  5. extreme problems It should be noted that the numerals 1-5 have no arithmetic properties and should not be used as a cardinal score. The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 100-'the best health you can imagine' and 0-'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.
Time Frame: 180 Days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidents of Adverse Events
Description: The number of subjects with AEs will be collected for each treatment group
Time Frame: 180 Days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Measurement of Local Tolerability
Description: Local tolerability will be assessed on a 0-3 scale (none, mild, moderate, severe).
Time Frame: 180 Days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Clinical Laboratory Evaluations
Description: The number of subjects with clinical laboratory values categorized as below (vital signs, 12 lead electrocardiogram, Physical Exam), within, or above normal ranges will be evaluated (changes from baseline for each clinical laboratory parameter by treatment group and by study visit).
Time Frame: 180 Days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Measurement of Vital Signs
Description: Blood pressure (systolic blood pressure [SBP], diastolic blood pressure [DBP] and pulse will be measured. Measurement of actual values and changes from baseline will be calculated. Vital signs The number of subjects with vital signs values categorized as below, within, or above normal ranges (change from baseline for each parameter by period, by treatment group and by study visit).
Time Frame: 180 Days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Measurement of 12-lead ECG Readings
Description: The number of subjects with normal and abnormal ECG findings will be measured for each treatment group at each time point for QT and the QT interval corrected for heart rate (QTc) calculated using Fridericia's QT correction methods.
Time Frame: 180 Days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Physical Examination Findings
Description: The number of subjects with normal and abnormal findings in the complete physical examination for each treatment group. This is a limited physical examination to include HEENT, cardiorespiratory, abdomen, and range of motion.
Time Frame: 180 Days
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Measurement of Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Measurement of the extent of absorption using estimates of the area-under-the-curve (AUC).
Time Frame: 180 Days
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Measurement of Peak Plasma Concentration (Cmax)
Description: Measurement of therate-of-absorption using the maximum concentration (Cmax) and the time of Cmax (Tmax).
Time Frame: 180 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The maximum study duration for each subject was approximately 291 days.
Arm/Group | CD5789 Cream 200 µg/g | CD5789 Cream 100 µg/g | CD5789 Cream Vehicle
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 10/23 | 7/21 | 11/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 Cream 200 µg/g (N=23) | CD5789 Cream 100 µg/g (N=21) | CD5789 Cream Vehicle (N=21)
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Dermatophytosis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Application site pain (General disorders) | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Feeling abnormal (General disorders) | 1 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03738800/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03738800/SAP_001.pdf